CLINICAL TRIAL: NCT04564911
Title: GLucose Monitoring Programme SingaporE, Phase 2(GLiMPSE2)
Brief Title: GLucose Monitoring Programme SingaporE, Phase 2 (GLiMPSE2)
Acronym: GLiMPSE2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Singapore General Hospital (Other)
Collaborators: National University Hospital, Singapore (Other); SingHealth Polyclinics (Other); National Healthcare Group Polyclinics (Other Government); National University Polyclinics, Singapore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GLiMPSE2
Record Dates: First submitted 2020-09-10; First posted 2020-09-25 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Diabetes Mellitus, Type 2; Flash Glucose Monitoring
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Flash Glucose Monitoring and Education (Experimental): Participants randomised to the experimental arm will receive an education package and wear the flash glucose monitoring system. They will use sensor glucose data for self-management.
  Interventions: Combination Product: Flash Glucose Monitoring and Education
- Capillary Glucose Monitoring and Education (Active Comparator): Participants randomised to the control arm will receive an education package and self-manage their glucose levels utilising a standard capillary blood glucose device, and keeping a glucose diary for the duration of the intervention period.
  Interventions: Combination Product: Capillary glucose monitoring and Education

INTERVENTIONS:
Combination Product: Flash Glucose Monitoring and Education — Participants will wear the flash glucose monitoring system, and receive an education package on how to self-manage their glucose levels. They will use the flash glucose monitoring system continuously for 6 weeks. From week 6 to week 24, the frequency of use of flash glucose monitoring will be reduced to one sensor every 4 weeks. They will receive education at weeks 0, 2, 8 and 16. They will also wear a blinded sensor for the last 2 weeks of the intervention period (week 25 to week 26). After the first 24 weeks, participants enter the observation phase (weeks 38 to 52) wherein they will be encouraged to continue monitoring their glucose levels through capillary glucose monitoring, during pre-meals and bedtime daily.
  Arms: Flash Glucose Monitoring and Education
Combination Product: Capillary glucose monitoring and Education — Participants will use a capillary glucose meter and receive an education package on how to self-manage their glucose levels. Participants will be encouraged to test their blood glucose levels at least twice a day, but preferably 4 times daily: pre-meal and bedtime blood glucose levels. They will receive education at weeks 0, 2, 8 and 16. They will wear a blinded sensor again after the last 2 weeks of the intervention period (week 24 to week 26). After the first 24 weeks, participants enter the observation phase (weeks 38 to 52) wherein they will be encouraged to continue monitoring their glucose levels through capillary glucose monitoring, during pre-meals and bedtime daily.
  Arms: Capillary Glucose Monitoring and Education

SUMMARY:
Many with type 2 diabetes (T2D) remain sub-optimally controlled. Structured programmes requiring dietary and lifestyle intervention have been shown to improve control but are time-and labour-intensive. The role for self-monitoring of blood glucose with capillary blood glucose (CBG) readings is uncertain. The use of flash glucose monitoring (FGM) with education may effect improvements in awareness and self-management behaviour and hence glycaemic control.

The investigators aim to compare the effects of FGM versus CBG fingersticks in the context of a structured education programme over a 6-month period in adults with type 2 diabetes. 200 adults (>21y) with sub-optimally controlled T2D (7.5-10%) on either diet-controlled, oral glucose lowering drugs or background insulin will be enrolled and randomised into the intervention arm (FGM and education) or control arm (capillary glucose fingersticks and education). The intervention arm will monitor glucose using FGM continuously for 6 weeks and intermittently thereafter up to 24 weeks. The control group will monitor glucose using CBG fingersticks up to 24 weeks. During the intervention period(0-24w), both arms will undergo the same schedule of visits (-2w, 0w, 8w, 16w, 24w) and 6 education sessions. Both groups will be followed up at weeks 38 and 52. Primary outcome is HbA1c change from baseline at 24 weeks. This study will provide novel data on the use of FGM versus CBG in Type 2 diabetes and its impact on glycaemic control.

DETAILED DESCRIPTION:
Up to 200 adults will be recruited from 5 different sites in Singapore. Following screening, consent and enrolment, all participants wear a blinded flash glucose monitoring system that is masked to the user and asked to continue testing capillary glucose readings at least once daily for 2 weeks (week -2 to week -1).Participants who are able to wear the sensor for the 2 weeks, and are monitoring capillary glucose levels at least 70% of the time for the 2 weeks (≥10 readings/2weeks), will carry on to be randomised to intervention or control group (week 0).

Upon fulfilling the criteria of blinded sensor wear of 2 weeks and 70% capillary glucose monitoring over 2 weeks, participants will be randomised into the control or the intervention arm, using web- based retrieval of randomisation allocation.

At baseline (week 0), all participants in both groups will receive baseline education on diabetes self-management, including blood glucose targets, role and timing of diabetes medications, and individualised education on macronutrient composition of meals and the goals of nutritional therapy in type 2 diabetes. Both groups will use the blinded FGM data at baseline for education. In total, both groups will receive 6 education sessions over the 24 week period, delivered by diabetes nurse educators or nurses and dietitians. The diabetes educators and physicians will be aligned towards a standardised curriculum for consistency of education through a train-the-trainer workshop.

Participants randomised to the control arm will receive an education package and be given education on how to self-manage glucose levels using a standard capillary blood glucose device. They will be encouraged to test blood glucose readings at least twice a day but preferably 4 times daily. Participants randomised to the intervention arm will wear the flash glucose monitoring system, and will be given education on how to use sensor glucose data for self-management. Flash glucose monitoring will be used continuously for 6 weeks. From week 6 to week 24, the frequency of use of flash glucose monitoring will be reduced to one sensor every 4 weeks.

The intervention period is for 24 weeks, followed by an observation period up to 52 weeks. After the 24-week intervention period, participants from both arms will wear a blinded sensor for the last 2 weeks of the intervention period (week 25 to week 26). During the observation period (weeks 24 to 52), participants in both arms will be encouraged to continue monitoring glucose levels.

Medication titrations will be left to the discretion of the primary physician. Physician consults will be at weeks 0, 8, 24, 38, 52. There will be no medication up-titration at week 0 although the physician may choose to optimize medications if needed: e.g. moving basal from bedtime to the morning to reduce the risk of nocturnal hypoglycemia or switching from a sulphonylurea agent to an alternative oral medication to reduce the risk of hypoglycaemia. If down-titration of medications is required, the reduction/cessation of sulphonylurea agents or insulin therapy will be encouraged to alleviate the risk of hypoglycaemia and promote weight loss. If there is no improvement in glycemic control or deterioration of glycaemic control at weeks 8 and 16 (laboratory HbA1c more than of equal to 8.5% for consecutive readings, one laboratory HbA1c more than or equal to 10% or a 2% point HbA1c increase from previous visit), medications may be up-titrated. The use of agents which do not increase the risk of hypoglycaemia and promote weight loss will be encouraged. If prandial insulin or premixed insulin is added to the treatment regimen from week 8 onwards, subjects will still remain within the study and be included in the analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (Age >21 years) with Type 2 diabetes (HbA1c 7.5 to 10% for 2 consecutive readings over the preceding 9 months at time of enrolment)
2. Singapore Citizen or Permanent Resident
3. Treatment with diet and exercise alone or other glucose-lowering therapies except prandial insulin. GLP-1 agonists and / or basal insulin (NPH insulin, Insulin Lantus, Insulin Toujeo, Insulin Detemir) are permitted.
4. Self-reported regular blood glucose testing via CBG (more than 3/week)

Exclusion Criteria:

1. Age above 75 years
2. Type 1 diabetes, monogenic diabetes
3. Prandial insulin (quick-acting insulin or premixed insulin)
4. Cancer requiring treatment in the past 5 years
5. Chronic renal failure (eGFR<45ml/min) or dialysis
6. Amputation of lower limbs (excluding toe amputations)
7. Bariatric surgery for weight loss
8. Current systemic treatment with steroids
9. Pregnancy, attempting pregnancy or lactation.
10. Haemolytic anaemia or haemoglobinopathy
11. Prior use of the flash glucose monitoring system for more than 3 times

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2020-12-22 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline HbA1c at week 24 | 24 weeks
  Measurement of HbA1c will be performed at weeks 0 and 24

SECONDARY OUTCOMES:
Change from baseline Time in Range at week 26 | 26 weeks
  Measurement of glucose indices will be done using Pro sensor at weeks 0 and 25-26, expressed as percentage of a day
Change in Baseline % Time Below Range at week 26 | 26 weeks
  Measurement of glucose indices will be done using Pro sensor at weeks 0 and 25-26, expressed as percentage of a day
Change from baseline % CV glucose at week 26 | 26 weeks
  Expressed as %CV glucose (standard deviation/ mean glucose), from pro sensor data at week 25-26
Change in Weight from baseline at week 24 | 24 weeks
  Anthropometry will be performed at weeks 24, expressed in kg
Change in Body Mass Index from baseline at week 24 | 24 weeks
  Anthropometry will be performed at weeks 24, expressed as kg/m2
Change in both systolic and diastolic blood pressure from baseline at week 24 | 24 weeks
  Expressed in mmHg
Change in score from baseline using the Work productivity and daily activity impairment questionnaire | 24 weeks
  Expressed as impairment percentages (0-100%), with higher scores indicating greater impairment and less productivity
Change from baseline in Diabetes Distress Scale score | 24 weeks
  Expressed as a mean score (sum of each score on the scale divided by the number of items on the score), a higher score (>3) indicating higher level of diabetes related distress
Change from baseline in EuroQol-5D-5L (5 level) utilities score. | 24 weeks
  The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The second part of the questionnaire consists of a visual analogue scale (VAS) on which the patient rates his/her perceived health from 0 (the worst imaginable health) to 100 (the best imaginable health). The EuroQol-5D-5L index will be calculated through comparison with a Singapore value set, with a higher score indicating a better health state utility.
Qualitative questionnaire | 24 weeks
  Questionnaire to assess the acceptability of the wear of the flash glucose monitoring system (experimental arm only)
Number of individuals requiring medication up-titration from baseline to week 24 | 24 weeks
  Number of additional oral medications added since baseline visit including addition of insulin

CONTACTS AND LOCATIONS:
Overall Officials: Daphne SL Gardner, MD, Principal Investigator — Singapore General Hospital
Locations (3):
- Singapore (3):
  - Pasir Ris Polyclinic, Singapore
  - National Healthcare Group, Singapore
  - National University Hospital, Singapore

IPD SHARING:
Plan to Share IPD: No